CLINICAL TRIAL: NCT02408432
Title: Intravenous Administration of Allogeneic Bone Marrow Derived Multipotent Mesenchymal Stromal Cells (MSCs) in Patients With Recent Onset Anthracycline-Associated Cardiomyopathy
Brief Title: Bone Marrow Derived Mesenchymal Stem Cells in Improving Heart Function in Patients With Heart Failure Caused by Anthracyclines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0519; NCI-2015-00969 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0519 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Cardiomyopathy; Heart Failure
MeSH Terms: conditions — Cardiomyopathies; Heart Failure | interventions — Standard of Care; Mesenchymal Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (hMSCs) (Experimental): Patients receive allogeneic hMSCs IV over 10-20 minutes once weekly for 4 weeks and standard of care drugs for heart failure.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Standard of Care; Drug: Mesenchymal Stem Cell Transplantation
- Arm II (standard of care drugs) (Active Comparator): Patients receive only standard of care drugs for heart failure.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Standard of Care; Drug: Mesenchymal Stem Cell Transplantation

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Standard of Care — Undergo mesenchymal stem cell infusion
Drug: Mesenchymal Stem Cell Transplantation — Undergo mesenchymal stem cell infusion

SUMMARY:
This randomized pilot phase I trial studies the side effects and best method of delivery of bone marrow derived mesenchymal stem cells (MSCs) in improving heart function in patients with heart failure caused by anthracyclines (a type of chemotherapy drug used in cancer treatment). MSCs are a type of stem cell that can be removed from bone marrow and grown into many different cell types that can be used to treat cancer and other diseases, such as heart failure. Bone marrow derived MSCs may promote heart muscle cells repair and lead to reverse remodeling and ultimately improve heart function and decrease morbidity and mortality from progression to advanced heart failure.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To demonstrate the safety of allogeneic human mesenchymal stem cells (hMSCs) administered by intravenous infusion in patients with left ventricular (LV) dysfunction and heart failure secondary to chemotherapy with anthracyclines.

SECONDARY OBJECTIVE:

I. To demonstrate the efficacy of allogeneic hMSCs administered by intravenous infusion in patients with left ventricular dysfunction (left ventricular ejection fraction [LVEF] < 40%) and heart failure secondary to treatment with anthracyclines.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive allogeneic hMSCs intravenously (IV) over 10-20 minutes once weekly for 4 weeks and standard of care drugs for heart failure.

ARM II: Patients receive only standard of care drugs for heart failure.

After completion of study treatment, patients are followed up monthly for 6 months and then at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with LVEF =< 40% from treatment with anthracyclines for all malignancies at any dose at any time without evidence of other causes of cardiomyopathy
* Documented New York Heart Association (NYHA) class I, II and III
* Been treated with appropriate maximal medical therapy for heart failure
* Able to perform 6 minute walk test
* Patient or legally authorized representative able to sign informed consent
* Patients with persistent LV dysfunction 90 days after discontinuation of trastuzumab

Exclusion Criteria:

* Evidence of ischemic heart disease as determined by study cardiologist
* Significant valvular disease; (aortic stenosis [AS] with aortic valve area [AVA] < 1.5 and severe aortic regurgitation [AR] and mitral regurgitation [MR])
* History of familial cardiomyopathy
* Recent documented myocarditis within 2 months of consent
* History of infiltrative cardiomyopathy or restrictive cardiomyopathy
* Epidermal growth factor receptor (eGFR) < 50 by Mayo or Cockcroft formula
* Liver function tests > 3 x upper limit of normal
* NYHA class IV heart failure
* Inotropic dependence
* Unstable or life-threatening arrhythmia
* Coagulopathy international normalized ratio (INR) > 1.5
* Mechanical or bioprosthetic heart valve
* Cardiogenic shock
* Breast feeding and/or pregnant women
* Autoimmune disorders on current immunosuppressive therapy
* Active infection not responding to appropriate therapy as determined by study chair
* Trastuzumab treatment within the last 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events of intravenous injection of human mesenchymal stem cells (hMSCs) in patients with recent onset left ventricular systolic dysfunction from anthracyclines | Up to 6 months
  Statistical analyses of safety will be descriptive. In particular, will provide a table of adverse events.

SECONDARY OUTCOMES:
Change in improvement in left ventricular systolic function by 7 points | Baseline up to 6 months
  Change from baseline left ventricular ejection fraction (LVEF) at 6 months after randomization, expressed as a percentage. The comparison will be between the two groups of patients.
Development of acute heart failure decompensation | Up to 6 months
  As regards statistical analyses, the results of the trial will be displayed in table format. Will provide confidence intervals of the differences in change from baseline between investigational and control groups. These intervals and the associate p-values will be calculated using two-sample t-tests, with no adjustments for multiple comparisons.
Emergency center visits for heart failure | Up to 6 months
  As regards statistical analyses, the results of the trial will be displayed in table format. Will provide confidence intervals of the differences in change from baseline between investigational and control groups. These intervals and the associate p-values will be calculated using two-sample t-tests, with no adjustments for multiple comparisons.
Need for new pacemaker/automatic implantable cardioverter defibrillator | Up to 6 months
  As regards statistical analyses, the results of the trial will be displayed in table format. Will provide confidence intervals of the differences in change from baseline between investigational and control groups. These intervals and the associate p-values will be calculated using two-sample t-tests, with no adjustments for multiple comparisons.
New onset arrhythmias | Up to 6 months
  As regards statistical analyses, the results of the trial will be displayed in table format. Will provide confidence intervals of the differences in change from baseline between investigational and control groups. These intervals and the associate p-values will be calculated using two-sample t-tests, with no adjustments for multiple comparisons.
Sudden cardiac death | Up to 6 months
  As regards statistical analyses, the results of the trial will be displayed in table format. Will provide confidence intervals of the differences in change from baseline between investigational and control groups. These intervals and the associate p-values will be calculated using two-sample t-tests, with no adjustments for multiple comparisons.
Acute pulmonary edema | Up to 6 months
  As regards statistical analyses, the results of the trial will be displayed in table format. Will provide confidence intervals of the differences in change from baseline between investigational and control groups. These intervals and the associate p-values will be calculated using two-sample t-tests, with no adjustments for multiple comparisons.
Asymptomatic decrease in left ventricular ejection fraction (LVEF) of > 10% | Baseline to up to 6 months
  As regards statistical analyses, the results of the trial will be displayed in table format. Will provide confidence intervals of the differences in change from baseline between investigational and control groups. These intervals and the associate p-values will be calculated using two-sample t-tests, with no adjustments for multiple comparisons.
Heart failure admission | Up to 6 months
  As regards statistical analyses, the results of the trial will be displayed in table format. Will provide confidence intervals of the differences in change from baseline between investigational and control groups. These intervals and the associate p-values will be calculated using two-sample t-tests, with no adjustments for multiple comparisons.
Progression free survival | Up to 12 months
  As regards statistical analyses, the results of the trial will be displayed in table format. Will provide confidence intervals of the differences in change from baseline between investigational and control groups. These intervals and the associate p-values will be calculated using two-sample t-tests, with no adjustments for multiple comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Olson, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org